CLINICAL TRIAL: NCT03774641
Title: A Pilot Study of Prophylactic Management of Lamotrigine for Bipolar Disorder in Pregnant Women
Brief Title: A Pilot Study of Prophylactic Management of Lamotrigine in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00162134; 1R01AG058671 (NIH)
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Disorder; Major Depressive Disorder; Schizo Affective Disorder
Keywords: Lamotrigine; Bipolar Disorder; Major Depressive Disorder; Schizo Affective Disorder
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Psychotic Disorders | interventions — Lamotrigine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Taking Lamotrigine: Lamotrigine (Lamictal), dosage will be based on a reference concentration of blood-serum levels
  Interventions: Drug: Lamictal

INTERVENTIONS:
Drug: Lamictal — Blood-serum levels will be checked monthly during pregnancy and reference concentration will be maintained
  Other Names: Lamotrigine

SUMMARY:
Pregnant women who are taking lamotrigine will be evaluated monthly during pregnancy including a clinical evaluation and a blood draw for lamotrigine levels at each visit. Based on the Therapeutic Drug Monitoring protocol, participant's lamotrigine dosing will be adjusted as needed based on participant's blood levels compared to the reference concentration that was obtained prior to pregnancy or early in pregnancy while clinically stable. After delivery participant and participant's infants will be assessed for mood and functioning at 1, 2, 4, and 6 weeks postpartum.

DETAILED DESCRIPTION:
Studies have demonstrated that at least 80% of women who stop mood stabilizing medications for pregnancy relapse psychiatrically. However, relapse is also quite common in women who continue taking mood stabilizing medication with studies demonstrating approximately a 30-37% relapse rate-most with depressive episodes. One likely explanation for the high relapse rate of Bipolar Disorder during pregnancy despite continued mood stabilizing medication is decreasing blood levels of mood stabilizing medications during the course of pregnancy. Pregnancy induces both pharmacokinetic and pharmacodynamic changes, which can result in decreased serum blood levels and decreased treatment efficacy. Therapeutic drug monitoring is considered standard of care for a number of psychiatric medications. Therapeutic drug monitoring can be an especially crucial guide to clinical treatment during pregnancy, but remarkably, there are no established protocols for the monitoring of levels and dosing of psychiatric medications in pregnancy. Most pregnant psychiatric patients are therefore managed based on symptom recurrence. In contrast, there are established protocols for monitoring blood levels and prophylactic management of antiepileptic medications for epilepsy, including lamotrigine which is also a mood stabilizing medication. The investigators will collect pilot data on the psychiatric outcomes, adverse events, and obstetrical and infant outcomes of pregnant women with Bipolar Disorder who undergo prophylactic therapeutic drug monitoring for a commonly used mood stabilizing medication during pregnancy- lamotrigine. In the epilepsy literature, there is a published protocol for lamotrigine management before, during, and after pregnancy for seizure control; the investigators will use this protocol as a guide.

ELIGIBILITY:
Inclusion Criteria:

* pregnant, prior or 20 weeks
* currently taking Lamotrigine and plan to continue throughout pregnancy
* history of Bipolar Disorder, Major Depressive Disorder, Schizoaffective Disorder or other psychiatric illness, currently stable
* may be taking other psychiatric medications

Exclusion Criteria:

* suicidal/clinically unstable
* alcohol, marijuana, or other drug dependence in last 90 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who are currently taking Lamotrigine for Bipolar Disorder, Major Depressive Disorder, Schizoaffective Disorder, or another psychiatric illness, and plan to continue throughout pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Change in Mood as assessed by The Edinburgh Postnatal Rating Scale | Monthly, after enrollment, up to 10 months
  Self-reported experience of depressive symptoms over the past 7 days, each item is scored 0-3 (0=not experiencing the symptom, 3=experiencing the symptom most of the time) yielding a total between 0 and 30. A score of 0-9 indicates little to no depressive symptoms and a score from 10-30 indicates significant depressive symptoms.
Change in Mood as assessed by The Young Mania Rating Scale | Monthly, after enrollment, up to 10 months
  Clinical interview that measures manic symptoms in the past 2 weeks, each item is scored 0-4 (0=absent, 4=fully present) yielding a total between 0 and 44. Any score above 0 indicates a possible manic episode.
Side Effect as assessed by the Udvalg for Kliniske Undersøgelser Side Effects Rating Scale | Monthly, after enrollment, up to 10 months
  Clinical interview that measures current, or in the past 72 hours, side effects of medication, each item is scored 0-3 (0=not or doubtfully present, 3=severe), yielding a total between 0 and 168. Any score above 0 indicates a possible causal relationship between medication and side effects.
Side Effect as assessed by the Frequency, Intensity, and Burden of Side Effects Rating Scale | Monthly, after enrollment, up to 10 months
  Self-reported frequency, intensity, and burden of side effects in the past week, each item is scored 0-6 (0=no side effects/impairment, 6=present all the time/intolerable/unable to function) yielding a total between 0 and 18. For each item, a score of 0-2 indicates treatment should continue, a score of 3-4 indicates the side effect should be addressed, and a score of 5-6 indicates a change in treatment is needed.
Change in Infant Habituation as assessed by the Neonatal Intensive Care Unit Network Neurobehavioral Scale | At 1, 2, 4, and 6 weeks postpartum
  Neurobehavioral assessment measuring infant's ability to shut down response to a stimulus, the item is scored 1-9, a low score indicates no decrement in response over 10 stimuli and a high score indicates a shut down of response after 1-2 stimuli
Change in Infant Attention as assessed by the Neonatal Intensive Care Unit Network Neurobehavioral Scale | At 1, 2, 4, and 6 weeks postpartum
  Neurobehavioral assessment measuring infant's response to a stimulus, the item is scored 1-9, a low score indicates no response and a high score indicates alerting to stimulus
Change in Infant Self-Regulation as assessed by the Neonatal Intensive Care Unit Network Neurobehavioral Scale | At 1, 2, 4, and 6 weeks postpartum
  Neurobehavioral assessment measuring infant's ability to self-regulate, the item is scored 1-9, a low score indicates the infant makes no attempt to quiet self and a high score indicates the infant consistently quiets self for sustained periods
Change in Infant Arousal as assessed by the Neonatal Intensive Care Unit Network Neurobehavioral Scale | At 1, 2, 4, and 6 weeks postpartum
  Neurobehavioral assessment measuring infant's arousal, the item is scored 1-9, a low score indicates a low level of arousal to all stimuli and a high score indicates the infant achieves insulated crying
Change in Infant Tonicity as assessed by the Neonatal Intensive Care Unit Network Neurobehavioral Scale | At 1, 2, 4, and 6 weeks postpartum
  Neurobehavioral assessment measuring infant's body tone, the item is scored 1-9, a low score indicates the infant is flaccid and a high score indicates the infant is hypertonic
Change in Infant Reflexes as assessed by the Neonatal Intensive Care Unit Network Neurobehavioral Scale | At 1, 2, 4, and 6 weeks postpartum
  Neurobehavioral assessment measuring infant's reflexes, the item is scored 1-5, a low score indicates no response and a high score indicates a strong response
Change in Infant Quality of Movement as assessed by the Neonatal Intensive Care Unit Network Neurobehavioral Scale | At 1, 2, 4, and 6 weeks postpartum
  Neurobehavioral assessment measuring infant's power and flexibility, the item is scored 1-5, a low score indicates no resistance/movement and a high score indicates strong resistance/movement
Gestational Age at Birth in Weeks assessed by Review of the Infant Delivery Chart | At 2 weeks postpartum visit, up to 15 minutes
Birth Length in Inches assessed by Review of the Infant Delivery Chart | At 2 weeks postpartum visit, up to 15 minutes
Birth Weight in pounds assessed by Review of the Infant Delivery Chart | At 2 weeks postpartum visit, up to 15 minutes
APGAR Score at 1 Minute assessed by Review of the Infant Delivery Chart | At 2 weeks postpartum visit, up to 15 minutes
APGAR Score at 5 Minutes assessed by Review of the Infant Delivery Chart | At 2 weeks postpartum visit, up to 15 minutes
Assessment of Neonatal Intensive Care Unit Admission by Review of the Infant Delivery Chart | At 2 weeks postpartum visit, up to 15 minutes
  By reviewing the infant delivery chart, the outcome will be "yes" if the infant was admitted to the Neonatal Intensive Care Unit and "no" if the infant was not admitted

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Standeven, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- 550 N Broadway, Baltimore, Maryland, United States

REFERENCES:
- [Background] Viguera AC, Whitfield T, Baldessarini RJ, Newport DJ, Stowe Z, Reminick A, Zurick A, Cohen LS. Risk of recurrence in women with bipolar disorder during pregnancy: prospective study of mood stabilizer discontinuation. Am J Psychiatry. 2007 Dec;164(12):1817-24; quiz 1923. doi: 10.1176/appi.ajp.2007.06101639. PMID 18056236
- [Background] Newport DJ, Stowe ZN, Viguera AC, Calamaras MR, Juric S, Knight B, Pennell PB, Baldessarini RJ. Lamotrigine in bipolar disorder: efficacy during pregnancy. Bipolar Disord. 2008 May;10(3):432-6. doi: 10.1111/j.1399-5618.2007.00565.x. PMID 18402631
- [Background] Le Strat Y, Dubertret C, Le Foll B. Prevalence and correlates of major depressive episode in pregnant and postpartum women in the United States. J Affect Disord. 2011 Dec;135(1-3):128-38. doi: 10.1016/j.jad.2011.07.004. Epub 2011 Jul 29. PMID 21802737
- [Background] Barker ED, Kirkham N, Ng J, Jensen SK. Prenatal maternal depression symptoms and nutrition, and child cognitive function. Br J Psychiatry. 2013 Dec;203(6):417-21. doi: 10.1192/bjp.bp.113.129486. Epub 2013 Oct 10. PMID 24115347
- [Background] McPhie S, Skouteris H, Fuller-Tyszkiewicz M, Hill B, Jacka F, O'Neil A. Relationships between mental health symptoms and body mass index in women with and without excessive weight gain during pregnancy. Midwifery. 2015 Jan;31(1):138-46. doi: 10.1016/j.midw.2014.07.004. Epub 2014 Jul 19. PMID 25086989
- [Background] Kim HG, Mandell M, Crandall C, Kuskowski MA, Dieperink B, Buchberger RL. Antenatal psychiatric illness and adequacy of prenatal care in an ethnically diverse inner-city obstetric population. Arch Womens Ment Health. 2006 Mar;9(2):103-7. doi: 10.1007/s00737-005-0117-5. Epub 2005 Dec 29. PMID 16380813
- [Background] Grigoriadis S, VonderPorten EH, Mamisashvili L, Tomlinson G, Dennis CL, Koren G, Steiner M, Mousmanis P, Cheung A, Radford K, Martinovic J, Ross LE. The impact of maternal depression during pregnancy on perinatal outcomes: a systematic review and meta-analysis. J Clin Psychiatry. 2013 Apr;74(4):e321-41. doi: 10.4088/JCP.12r07968. PMID 23656857
- [Background] Dennis CL, McQueen K. The relationship between infant-feeding outcomes and postpartum depression: a qualitative systematic review. Pediatrics. 2009 Apr;123(4):e736-51. doi: 10.1542/peds.2008-1629. PMID 19336362
- [Background] Diego MA, Field T, Hernandez-Reif M, Cullen C, Schanberg S, Kuhn C. Prepartum, postpartum, and chronic depression effects on newborns. Psychiatry. 2004 Spring;67(1):63-80. doi: 10.1521/psyc.67.1.63.31251. PMID 15139586
- [Background] Ashman SB, Dawson G, Panagiotides H, Yamada E, Wilkinson CW. Stress hormone levels of children of depressed mothers. Dev Psychopathol. 2002 Spring;14(2):333-49. doi: 10.1017/s0954579402002080. PMID 12030695
- [Background] Essex MJ, Klein MH, Cho E, Kalin NH. Maternal stress beginning in infancy may sensitize children to later stress exposure: effects on cortisol and behavior. Biol Psychiatry. 2002 Oct 15;52(8):776-84. doi: 10.1016/s0006-3223(02)01553-6. PMID 12372649
- [Background] Halligan SL, Herbert J, Goodyer IM, Murray L. Exposure to postnatal depression predicts elevated cortisol in adolescent offspring. Biol Psychiatry. 2004 Feb 15;55(4):376-81. doi: 10.1016/j.biopsych.2003.09.013. PMID 14960290
- [Background] Robertson E, Grace S, Wallington T, Stewart DE. Antenatal risk factors for postpartum depression: a synthesis of recent literature. Gen Hosp Psychiatry. 2004 Jul-Aug;26(4):289-95. doi: 10.1016/j.genhosppsych.2004.02.006. PMID 15234824
- [Background] Akman I, Kuscu K, Ozdemir N, Yurdakul Z, Solakoglu M, Orhan L, Karabekiroglu A, Ozek E. Mothers' postpartum psychological adjustment and infantile colic. Arch Dis Child. 2006 May;91(5):417-9. doi: 10.1136/adc.2005.083790. Epub 2006 Feb 1. PMID 16452109
- [Background] Flynn HA, Davis M, Marcus SM, Cunningham R, Blow FC. Rates of maternal depression in pediatric emergency department and relationship to child service utilization. Gen Hosp Psychiatry. 2004 Jul-Aug;26(4):316-22. doi: 10.1016/j.genhosppsych.2004.03.009. PMID 15234828
- [Background] McLearn KT, Minkovitz CS, Strobino DM, Marks E, Hou W. The timing of maternal depressive symptoms and mothers' parenting practices with young children: implications for pediatric practice. Pediatrics. 2006 Jul;118(1):e174-82. doi: 10.1542/peds.2005-1551. PMID 16818531
- [Background] Grace SL, Evindar A, Stewart DE. The effect of postpartum depression on child cognitive development and behavior: a review and critical analysis of the literature. Arch Womens Ment Health. 2003 Nov;6(4):263-74. doi: 10.1007/s00737-003-0024-6. PMID 14628179
- [Background] Deligiannidis KM, Byatt N, Freeman MP. Pharmacotherapy for mood disorders in pregnancy: a review of pharmacokinetic changes and clinical recommendations for therapeutic drug monitoring. J Clin Psychopharmacol. 2014 Apr;34(2):244-55. doi: 10.1097/JCP.0000000000000087. PMID 24525634
- [Background] Fotopoulou C, Kretz R, Bauer S, Schefold JC, Schmitz B, Dudenhausen JW, Henrich W. Prospectively assessed changes in lamotrigine-concentration in women with epilepsy during pregnancy, lactation and the neonatal period. Epilepsy Res. 2009 Jul;85(1):60-4. doi: 10.1016/j.eplepsyres.2009.02.011. Epub 2009 Mar 9. PMID 19272754
- [Background] Polepally AR, Pennell PB, Brundage RC, Stowe ZN, Newport DJ, Viguera AC, Ritchie JC, Birnbaum AK. MODEL-BASED LAMOTRIGINE CLEARANCE CHANGES DURING PREGNANCY: CLINICAL IMPLICATION. Ann Clin Transl Neurol. 2014 Feb;1(2):99-106. doi: 10.1002/acn3.29. PMID 24883336
- [Background] Hirsch LJ, Weintraub D, Du Y, Buchsbaum R, Spencer HT, Hager M, Straka T, Bazil CW, Adams DJ, Resor SR Jr, Morrell MJ. Correlating lamotrigine serum concentrations with tolerability in patients with epilepsy. Neurology. 2004 Sep 28;63(6):1022-6. doi: 10.1212/01.wnl.0000138424.33979.0c. PMID 15452293
- [Background] Sabers A. Algorithm for lamotrigine dose adjustment before, during, and after pregnancy. Acta Neurol Scand. 2012 Jul;126(1):e1-4. doi: 10.1111/j.1600-0404.2011.01627.x. Epub 2011 Dec 9. PMID 22150770
- [Background] Clark CT, Klein AM, Perel JM, Helsel J, Wisner KL. Lamotrigine dosing for pregnant patients with bipolar disorder. Am J Psychiatry. 2013 Nov;170(11):1240-7. doi: 10.1176/appi.ajp.2013.13010006. PMID 24185239

DOCUMENTS (1):
  • Study Protocol (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT03774641/Prot_000.pdf